CLINICAL TRIAL: NCT01135485
Title: Evaluation of Panel Reactive Antibody in Children Following Stage I Palliation for Hypoplastic Left Heart Syndrome
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 09-007242
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Study group I: Study group I will include children who have undergone stage I palliation employing allograft material for left ventricular outflow tract reconstruction at CHOP during infancy (<1 year of age). Stage I palliation is defined as an operation in which augmentation of the native ascending aorta and aortic arch is performed to bypass atresia or critical obstruction of the left heart structures.
- Study Group II: Study group II who have undergone stage II palliation in which allograft material is used, but have not undergone antecedent stage I palliation. Stage II palliation is defined as a superior cavopulmonary anastomosis in which the superior vena cava is anastomosed to the ipsilateral pulmonary artery via either the bidirectional Glenn or hemi-Fontan procedures.
- Control Group: The control group who have undergone palliative or corrective surgery for congenital heart disease during infancy (<1 year of age) not requiring allograft material.

SUMMARY:
The purpose of this study is to determine whether children and adolescents 8-18 years of age with HLHS and related lesions who have undergone stage I palliation during infancy using an allograft patch demonstrate continued evidence of HLA antibody formation.

DETAILED DESCRIPTION:
This study will be of a prospective cross-sectional design, consisting of three groups. The first two groups (study groups) will consist of (1) subjects with HLHS and other related lesions who have undergone stage I palliation using an allograft patch during infancy and (2) subjects with "single ventricle" lesions who have undergone stage II palliation using allograft without antecedent stage I palliation. The third group (control group) will consist of subjects who have undergone corrective or palliative surgery for CHD during infancy in which an allograft patch was not used, and in which there have been no further exposures to allograft. We have chosen to study both (1) subjects who have undergone stage I and II palliation and (2)subjects who have undergone stage II palliation only in an attempt to distinguish between sensitization that may occur from allograft exposure during stage I palliation and that which may occur during stage II palliation.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 8 and 18 years of age.
* Parents/guardian permission (informed consent)
* Assent of the study subject
* Subjects followed within the CHOP Cardiology Division
* Operative note(s) available for review in medical record
* Have undergone stage I, stage II palliation, or corrective surgery for congenital heart disease during infancy (<1 year of age) not requiring allograft material.

Exclusion Criteria:

* Refusal or withdrawal of informed consent and/or assent.
* unavailability of medical records to confirm operative details.
* Additional surgeries (e.g., other than stage I or II palliation) utilizing allograft
* Exposure to allograft at any point in control group AGE <8 or >18 years
* Presence of genetic syndrome known to affect immunologic function (e.g., DiGeorge syndrome)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents between 8 and 18 years of age
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary and Secondary Endpoints | 2 years
  The primary objective is to determine PRA in a cross-sectional analysis of children and adolescents who have undergone stage I palliation for HLHS and related lesions during infancy, and comparing PRA measurements in a similarly aged group of children and adolescents who have undergone congenital heart surgery during infancy without use of allograft.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Shaddy, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States